CLINICAL TRIAL: NCT00402389
Title: Randomized Controlled Trial of Omega-3 Fatty Acids for Perinatal Depression
Brief Title: Use of Omega-3 Fatty Acids for Perinatal Depression
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Arizona (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: K23MH066265 (NIH); K23MH066265 (NIH); DATR AK-TNAI2
Record Dates: First submitted 2006-11-20; First posted 2006-11-22 (Estimated); Last update posted 2013-03-29 (Estimated); Status verified 2013-03

CONDITIONS: Depression; Depression, Postpartum
Keywords: Perinatal Depression; Postpartum Depression; Omega-3 Fatty Acids; Eicosapentaenoic Acid (EPA); Docosahexaenoic Acid (DHA); Pregnancy; Psychotherapy
MeSH Terms: conditions — Depression; Depression, Postpartum | interventions — Fatty Acids, Omega-3

STUDY DESIGN:
Who Masked: Participant, Care Provider

ARMS (2):
- 1 (Experimental): Participants assigned to take omega-3 fatty acids
  Interventions: Drug: Omega-3 Fatty Acids (EPA plus DHA); Behavioral: Supportive psychotherapy
- 2 (Placebo Comparator): Participants assigned to take placebo
  Interventions: Behavioral: Supportive psychotherapy; Drug: Placebo

INTERVENTIONS:
Drug: Omega-3 Fatty Acids (EPA plus DHA) — Four capsules will be taken daily for 8 weeks.
  Arms: 1
Behavioral: Supportive psychotherapy — Supportive psychotherapy will provide education to increase understanding of the condition, guidance on how to cope with depression, and methods on how to improve self-esteem.
Drug: Placebo — Four capsules will be taken daily for 8 weeks.
  Arms: 2

SUMMARY:
This study will evaluate the effectiveness of using omega-3 fatty acids to treat women with perinatal depression.

DETAILED DESCRIPTION:
Depression is the chief cause of disease-associated disability in women. Because of the highs and lows during pregnancy through the first year of motherhood, expectant and new mothers are particularly prone to depression. Approximately 10% to 15% of women experience perinatal depression, which includes depression during pregnancy and/or postpartum depression. Signs of perinatal depression include persistent feelings of anxiety, guilt, or hopelessness; irregular sleep and appetite patterns; lethargy; disinterest in the infant or family activities; excessive irritability and restlessness; thoughts of hurting self or infant; inability to concentrate; and lack of enjoyment in previously enjoyed activities. Depression occurring during pregnancy and postpartum can have a negative impact on the development and health of the baby. Additionally, maternal stress in humans is associated with lower birth weights and lower gestational ages at birth. Currently, there is a lack of knowledge on the use of antidepressants during pregnancy and postpartum, making this a significant health issue. Earlier studies have suggested that a depletion of omega-3 fatty acids during pregnancy might be the cause of depression and mood disorders in pregnant women. This study will evaluate the effectiveness of using omega-3 fatty acids to treat women with perinatal depression.

Participation in this double-blind study will last about 9 weeks. All participants will attend an initial screening visit and subsequent study visits, which will occur bi-weekly throughout the treatment phase. During these visits, participants will be asked questions about their medical and substance use history, demographic information, and eating behaviors. Participants will also complete questionnaires and interviews that will be used to assess their mental status, depression levels, marital/partner satisfaction levels, social/functional abilities, and overall mood levels. After the initial screening visit, eligible participants will be randomly assigned to receive either omega-3 fatty acids or placebo capsules. Participants in each group will be required to take four capsules on a daily basis for 8 weeks. During this treatment phase, all participants will also attend six weekly 30-minute supportive psychotherapy sessions. Blood samples for omega-3 fatty acid analysis will be taken on the first and last visits.

ELIGIBILITY:
Inclusion Criteria:

* Women who are pregnant (12 to 32 weeks gestation) or postpartum
* Meets criteria for a major depressive episode
* Scores a minimum of 9 on the Edinburgh Postnatal Depression scale
* Must be able to be treated on an outpatient basis

Exclusion Criteria:

* Known intolerance or allergy to omega-3 fatty acid or fish oil
* Presently taking antidepressant medication
* Currently using heparin or warfarin (compounds used to prevent blood from clotting)
* Presence of psychotic symptoms
* History of mania (abnormally elevated mood state) or hypomania (same as mania but occurs at a much lesser degree)
* Active suicidal ideation (desire to commit suicide)

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 50 (Actual)
Dates: Start 2004-06; Primary Completion 2006-01 (Actual); Study Completion 2006-01 (Actual)

PRIMARY OUTCOMES:
Reduction of initial Edinburgh Postnatal Depression Scale (EPDS) score by 50% or more | Measured at Week 8
Reduction of EPDS score to less than or equal to 9 | Measured at Week 8
CGI change score achievement of "very much improved" or "much improved" | Measured at Week 8

SECONDARY OUTCOMES:
Significant reductions in outcome measures of functional status and reduction of SIGH-ADS score of 50% | Measured at Week 8
Changes in the level of omega-3 fatty acid composition of red blood cell membranes | Measured at Weeks 1 and 8

CONTACTS AND LOCATIONS:
Overall Officials: Marlene P. Freeman, MD, Principal Investigator — University of Arizona; Department of Psychiatry
Locations (1):
- Women's Mental Health Program; University of Arizona; Department of Psychiatry, Tucson, Arizona, United States

REFERENCES:
- [Result] Freeman MP, Hibbeln JR, Wisner KL, Brumbach BH, Watchman M, Gelenberg AJ. Randomized dose-ranging pilot trial of omega-3 fatty acids for postpartum depression. Acta Psychiatr Scand. 2006 Jan;113(1):31-5. doi: 10.1111/j.1600-0447.2005.00660.x. PMID 16390366